CLINICAL TRIAL: NCT01337778
Title: Empowering Daughters and Mother-in-laws to Mitigate Gender-based Violence and Promote Women's Health in India
Brief Title: Dil Mil (Hearts Together)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: St. John's Research Institute (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21HD062821-01A1 (NIH); 1R21HD062821-01A1 (NIH)
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Gender Based Violence; Women's Health
Keywords: gender based violence; maternal and child health; women; India
MeSH Terms: interventions — Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary Care for DILs (Active Comparator): Primary care for DILs will be offered based on national and international standards and include access to critical support services for women who have experienced gender-based violence. A comprehensive health examination for mothers-in-law will include a gynecological exam and screening for diabetes and hypertension, along with appropriate information, prescriptions, and/or referrals. We will routinely offer GBV-related resources, such as information, counseling, and referrals to all participants. Referrals will be documented using a Referral Care Form and reviewed on a routine basis to ensure that appropriate care is being provided and to detect any potential study-related risks.
  Interventions: Behavioral: Primary care for Daughters-in-Law
- Standard Care plus Dil Mil Intervention (Experimental): The Dil Mil intervention will be implemented during the second and third trimesters of the daughter-in-law's (DILs) pregnancy. It consists of 2 half-day group sessions with DILs, 5 half-day group sessions with mothers-in-law (MILs), and one joint half-day session with DILs and MILs. The sessions are based on participatory learning and action principles and use stories, role-play, and discussion to enhance participants' knowledge, skills, and social support. The DIL-MIL joint session ends in a short celebration (based on a traditional ritual) in which MILs bless their DILs, and the MIL sessions culminate in a ceremony in which MILs' position in the family and community is recognized and celebrated. MILs draw up a family health action plan and take a pledge to reduce gender-based violence (GBV) and protect and promote their family's health.
  Interventions: Behavioral: The Dil Mil Intervention

INTERVENTIONS:
Behavioral: Primary care for Daughters-in-Law — Primary care for DILs will be offered based on national and international standards and include access to critical support services for women who have experienced GBV.A comprehensive health examination for MILs will include a gynecological exam and screening for diabetes and hypertension, along with appropriate information, prescriptions, and/or referrals. We will routinely offer GBV-related resources, such as information, counseling, and referrals to all participants. Referrals will be documented using a Referral Care Form and reviewed on a routine basis to ensure that appropriate care is being provided and to detect any potential study-related risks.
  Arms: Primary Care for DILs
Behavioral: The Dil Mil Intervention — The Dil Mil intervention will be implemented during the second and third trimesters of the DILs' pregnancy. It consists of 2 half-day group sessions with DILs, 5 half-day group sessions with MILs, and one joint half-day session with DILs and MILs. The sessions are based on participatory learning and action principles and use stories, role-play, and discussion to enhance participants' knowledge, skills, and social support. Participants are encouraged to critically analyze their relationships and to develop and implement responses appropriate to their families and communities. The DIL-MIL joint session ends in a short celebration (based on a traditional ritual) in which MILs bless their DILs, and the MIL sessions culminate in a ceremony in which MILs' position in the family and community is recognized and celebrated. MILs draw up a family health action plan and take a pledge to reduce GBV and protect and promote their family's health.
  Arms: Standard Care plus Dil Mil Intervention

SUMMARY:
A growing body of research indicates that gender-based violence (GBV) is a major global public health challenge. Yet, there is a dearth of evidence to guide program planning and policy-making efforts to reduce GBV. Our study will evaluate the feasibility, safety, and potential effectiveness of an innovative women's empowerment intervention to reduce GBV and related adverse health outcomes. It is expected that the study findings will provide evidence to determine if a phase 3 effectiveness trial is merited and advance the science underlying GBV prevention.

DETAILED DESCRIPTION:
The prevalence of physical, psychological, and sexual gender-based violence (GBV) is staggeringly high among young, married women in India. However, few GBV prevention interventions have been implemented, and none of these interventions has been rigorously evaluated. The investigators aim to fill this gap by conducting exploratory research on an innovative women's empowerment-based GBV prevention intervention. The proposed study builds on our previous research in urban poor communities in Bangalore, India, which revealed that efforts to enhance young, married women's power and to mitigate GBV will be limited if the broader context of their lives, which is shaped mainly by the marital family, is unaddressed. Previous research suggests that mothers-in-law (MILs) are a strategic familial entry point and that it may be possible to redirect the power they wield in the family toward reducing GBV against daughters-in-law (DILs). Based on this evidence and women's empowerment approaches that have successfully reduced GBV elsewhere, the investigators developed the intervention Dil Mil (meaning "Hearts Together" in India's national language, Hindi).

Guided by the Social Cognitive Theory and Heise's social-ecological framework of GBV, Dil Mil aims to empower DIL-MIL dyads with knowledge, skills, and social support critical to the mitigation of GBV and related adverse health outcomes among DILs. The investigators chose antenatal care as the context for implementing this intervention because of women's nearly universal use of antenatal care in urban India. A phase 1 pilot study demonstrated that our approach is acceptable and likely to be safe. The aim of this R21 is to conduct a phase 2 trial to examine the feasibility, safety, and potential effectiveness of Dil Mil in order to determine if a phase 3 effectiveness trial is merited.

The proposed study is a randomized controlled trial with 140 dyads comprising pregnant DILs (aged 18 to 30 years, in their first or second trimester of pregnancy, with a history of GBV) and their MILs. Recruitment will take place at four primary health centers serving poor communities in Bangalore. Dyads will be offered standard care or standard care plus the Dil Mil intervention, and evaluations will be conducted at 3 months and 6 months postpartum. The investigators will characterize the study population using descriptive statistics and assess feasibility and safety of the intervention using qualitative and quantitative data (Aim 1). Data on the effect of the intervention on intermediary outcomes-the empowerment of DILs and MILs (Aim 2)-and on the incidence of GBV among DILs during the first 6 months postpartum, DILs' perceived quality of life and psychosocial status, and maternal and infant health outcomes (Aim 3) will be analyzed using the intention-to-treat principle. Based on this evidence, the investigators will determine if a phase 3 trial is merited. In conclusion, this study will generate important insights on a novel, urgently needed response to GBV in a high prevalence setting and is highly likely to have a significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

Daughters-in-Law:

* married
* age 18 years to 30 years
* have ever experienced physical, psychological, or sexual violence perpetrated by husbands, mothers-in-law, or other marital family members
* pregnant and in the first or second trimester
* Kannada or Tamil speaking
* able and willing to provide consent
* able and willing to refer their mother-in-law for study participation

Mothers-in-Law:

* Kannada or Tamil speaking
* able and willing to give informed consent to participate
* confirm that they are the mother-in-law of a daughter-in-law who is being recruited.

Exclusion Criteria:

* planning to move from the area before the daughter-in-law completes 6 months postpartum
* cognitively impaired
* major depression or dementia

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incident Gender-Based Violence (GBV) | 3 months postpartum
  Measured in terms of any physical, psychological, or sexual violence perpetrated by husbands, MILs, or other family members
Incident GBV | 6 months postpartum
  Measured in terms of any physical, psychological, or sexual violence perpetrated by husbands, MILs, or other family members

SECONDARY OUTCOMES:
Safety | 3 months postpartum
  Measured by the frequency of safety alerts and adverse events at enrollment and during the course of the study.
Safety | 6 months postpartum
  Measured by the frequency of safety alerts and adverse events at enrollment and during the course of the study.
Feasibility | 3 months postpartum
  Data on recruitment, adherence (in the intervention arm) and attrition rates will be examined
Feasibility | 6 months postpartum
  Data on recruitment, adherence (in the intervention arm) and attrition rates will be examined
Daughter-in-Laws' (DILs') Knowledge | 3 months postpartum
  DILs' knowledge about safety and the links between GBV and health, their gender-equitable attitudes, and their decision-making skills
DILs' Knowledge | 6 months postpartum
  DILs' knowledge about safety and the links between GBV and health, their gender-equitable attitudes, and their decision-making skills
Mother-in-Laws' Knowledge | 3 months postpartum
  MILs' knowledge about the links between GBV and health and their gender-equitable attitudes; and improved relationships between MILS and DILs measured in terms of enhanced social support and communication.
MILs' Knowledge | 6 months postpartum
  MILs' knowledge about the links between GBV and health and their gender-equitable attitudes; and improved relationships between MILS and DILs measured in terms of enhanced social support and communication.

CONTACTS AND LOCATIONS:
Overall Officials: Suneeta Krishnan, PhD, Principal Investigator — RTI International
Locations (1):
- St. John's Research Institute, St. John's National Academy of Health Sciences, Kormangala, Bangalore, India

REFERENCES:
- [Derived] Krishnan S, Subbiah K, Chandra P, Srinivasan K. Minimizing risks and monitoring safety of an antenatal care intervention to mitigate domestic violence among young Indian women: The Dil Mil trial. BMC Public Health. 2012 Nov 1;12:943. doi: 10.1186/1471-2458-12-943. PMID 23116189